CLINICAL TRIAL: NCT02505724
Title: Peer-coaching to Teach Faculty Surgeons an Advanced Laparoscopic Skill
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Vanessa Palter, Dr., Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 305-2013
Record Dates: First submitted 2015-07-20; First posted 2015-07-22 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Coaching; Technical Skill; Laparoscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional training (Active Comparator): Participants received access to a web-based tutorial for laparoscopic suturing and a box trainer for independent practice
  Interventions: Behavioral: conventional training
- Intervention (Experimental): Participants received access to a web-based tutorial for laparoscopic suturing and a box trainer for independent practice. In addition, they received two 1/2 hour peer-coaching sessions
  Interventions: Behavioral: peer-coaching

INTERVENTIONS:
Behavioral: conventional training — After completing the initial assessment, faculty randomized to the conventional training group received a link to a web-based instructional video. In addition, they were given a laparoscopic box trainer, laparoscopic instruments and sutures that they could use to practice with at their leisure.
  Arms: Conventional training
Behavioral: peer-coaching — Faculty randomized to the peer-coaching group received ½ hour of peer-coaching after completing the initial assessment on the simulator. Each faculty member sutured on the box trainer while being observed by his or her peer-coach. All study participants had the same peer-coach.After the coaching session, study participants received a link to the web-based video as well as the box trainer and supplies to independently practice laparoscopic suturing. Similar to individuals in the control group, no specific guidance regarding the amount of independent practice was given.
  Arms: Intervention

SUMMARY:
This single-blinded randomized controlled trial assesses the efficacy of peer-coaching to teach novice surgical faculty an advanced laparoscopic skill.

ELIGIBILITY:
Inclusion Criteria:

* surgical faculty in the division of general surgery or obstetrics and gynaecology.
* novices in laparoscopic suturing (performed <20 intra-corporeal stiches and knots)

Exclusion Criteria:

* n/a

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-07; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Technical Skill | Two weeks post intervention
  Technical skill as measured by the Objective Structured Assessment of Technical Skill (OSATS) global rating scale. Participants are scored on 4 domains from 0-5 (respect for tissue, precision of operative technique, economy of movements, confidence of movements). The maximum possible score is 20.